CLINICAL TRIAL: NCT06535789
Title: The Safety and Efficacy of Rapid Acting Inhaled Technosphere Insulin (Afrezza) Compared With Subcutaneous Insulin to Achieve Pregnancy-Specific Postprandial Targets Among Patients With Gestational Diabetes
Brief Title: Inhaled Insulin vs Rapid-acting Injections for Post-meal Glucose Control in Women With Gestational Diabetes
Acronym: INHALE-GDM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INHALE-GDM
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetes, Gestational; Pregnancy Complications; Glucose Metabolism Disorders; Glucose Intolerance During Pregnancy
Keywords: Gestational Diabetes; Inhaled Insulin
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Participants will complete two in-clinic meal sessions, with random assignment to receive either technosphere insulin (TI) or RAA insulin for the first meal and the other insulin for the second meal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- technosphere insulin (TI) (Experimental): All participants will ingest one standardized meal using technosphere insulin to manage their blood glucose
  Interventions: Drug: Inhaled Technosphere Insulin
- Rapid-acting insulin analog (No Intervention): All participants will ingest one standardized meal using their prescribed rapid-acting insulin analog (RAA) to manage their blood glucose

INTERVENTIONS:
Drug: Inhaled Technosphere Insulin — Patients will receive TI (Afrezza) to be compared to RAA following a breakfast meal
  Arms: technosphere insulin (TI)

SUMMARY:
Pregnant women aged 18-40 with gestational diabetes (GDM) will take part in this study. We want to see how two different insulin treatments affect their blood sugar after they eat. These women usually use a rapid-acting insulin analog (RAA) that's injected to control their blood sugar before and after meals. They will come to the clinic for two meal sessions. For the first meal, we will randomly decide if they will use the usual RAA insulin or a newer inhaled insulin called technosphere insulin (TI). They will use the other type of insulin for their second meal. After each meal, we will compare their blood sugar levels.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) affects up to 25% of births globally, and its rates continue to rise each year. Pregnancy is a dynamic time marked by rapid changes in physiology, anatomy, and metabolism that support the growth and development of the fetus. This period can also be vulnerable, as expectant mothers may experience shifts in body perception, food preferences, and physical fitness, which can lead to decreased self-esteem, depression, and anxiety. A diagnosis of GDM often catches women by surprise and may bring feelings of guilt and anxiety about the potential effects on their baby's health. For pregnant individuals unable to meet specific glucose targets through diet and exercise alone, insulin is recommended as the primary treatment. However, transitioning to insulin injections can provoke fear, stress, and discomfort-both emotionally and physically-for many patients. Consequently, some pregnant women opt for oral anti-diabetic medications like metformin or glyburide due to their apprehension about using insulin injections. Both of these drugs pass through the placenta and raise safety concerns, making them secondary choices according to the American Diabetes Association (ADA) and the American College of Obstetricians and Gynecologists (ACOG).

While GDM is typically managed with injectable insulin, inhalable insulin offers a potential alternative. Technosphere® Insulin inhalation powder (TI) is an ultra-rapid-acting insulin administered via oral inhalation using a breath-powered inhaler. It provides an alternative to injectable insulin for prandial glucose control. It consists of recombinant human insulin adsorbed onto fumaryl diketopiperazine (FDKP), a proprietary excipient that, at acidic pH, self-assembles into particles, and polysorbate 80. TI particles have a median diameter of approximately 2 to 2.5 μm, a size appropriate for inhalation into the lung. Following inhalation, Afrezza particles dissolve immediately at the physiologic pH of the lung, and insulin and FDKP are absorbed systemically. After administration of TI in adults, the maximum serum insulin concentration occurs in approximately 12 to 15 minutes (versus 45 to 60 minutes for RAA via subcutaneous route) and returns to near baseline levels in approximately 180 minutes (versus about 5 hours for RAA).

The United States Food and Drug Administration (FDA) approved TI Inhalation Powder and the Gen2 Inhaler (a dry powder device) as Afrezza® to improve blood sugar control in adults aged 18 years and older with diabetes on June 27, 2014. Inhaled TI has proven safe and effective in reducing postprandial (after-meal) hyperglycemia in individuals with Type 1 and Type 2 diabetes. It's important to note that TI units are not equivalent to injectable insulin units; TI's bioequivalent dose has been found to be about twice that of injectable rapid-acting insulin when prescribed for diabetes management.

All insulins, including TI, have a similar label wording with respect to use in pregnancy indicating that studies have not shown an association of insulin and birth defects and that there are risks to the mother and fetus associated with poorly controlled diabetes in pregnancy. Insulin, whether subcutaneously administered or inhaled, has not been demonstrated to cross the placenta secondary to its large molecular weight. TI's inert excipient FDKP is not metabolized and is fully excreted from the body with the majority in urine and some in the feces (i.e. for the amount swallowed). Animal studies using subcutaneous administration of carrier particles at 21 times human dosing demonstrated no adverse fertility, teratogenicity, or other developmental outcomes (described in Afrezza label).

TI's optimal dosing, efficacy and risk for hypoglycemia in pregnancy is unknown. Outside of pregnancy, TI has been shown to cause less hypoglycemia than RAA insulin. The dose conversions of TI from RAA therapy have not been characterized in pregnancy to effectively administer across gestation with the dynamic metabolic changes, although insulin resistance is high in the 3rd trimester and dosing is expected to be at least as high as in patients with T2D (~2X SQ insulin dosing).

The goal of this investigator-initiated randomized crossover trial is to assess the efficacy of TI in lowering PP glycemia and the frequency of hypoglycemia compared with subcutaneous RAA insulin among pregnant individuals with GDM.

ELIGIBILITY:
Inclusion Criteria

1. Ability to provide informed consent for study participation
2. Age ≥18 years and <41 years old
3. Singleton pregnancy at 24-34 weeks gestation
4. Diagnosis of GDM via standard 1-step or 2-step criteria
5. Treated with an insulin regimen that includes a RAA bolus of any type for breakfast, with a dose <20 units
6. Pre-pregnancy or first trimester body mass index (BMI) 25-45
7. Investigator believes that the protocol can be safely conducted by the participant
8. Able to read and speak English

Exclusion Criteria

1. Type 1 diabetes or type 2 diabetes
2. HbA1c ≥ 6.5%, FBG ≥125 mg/dl or 2-hr glucose ≥200 mg/dL on 75g OGTT, or random plasma glucose ≥200 mg/dL (consistent with pre-existing diabetes and not GDM diagnosis)
3. Current use of any non-insulin glucose lowering medication
4. Using TI (Afrezza), regular insulin, or ≥20 RAA units at breakfast (NPH is permissible)
5. Peak expiratory flow <80% predicted as measured by peak flow meter
6. Recent history of asthma (defined as using any medications to treat asthma within the last year), chronic obstructive pulmonary disease (COPD), or any other clinically important pulmonary disease (e.g., cystic fibrosis or bronchopulmonary dysplasia), or significant congenital or acquired cardiopulmonary disease as judged by the Investigator
7. Smoking (includes cigarettes, cigars, pipes, and/or vaping devices) within 90 days prior to screening
8. History or current diagnosis of lung cancer
9. Current or anticipated use of oral, inhaled or injectable glucocorticoids during the time period of the trial (topical glucocorticoid use is acceptable)
10. Renal or hepatic impairment that in the investigator's judgment poses a safety risk for the study participant
11. Recurrent Level 2 (blood glucose <54 mg/dL) or Level 3 severe hypoglycemia events
12. Current use of non-cardio-selective beta blockers
13. Being a member of the study team, having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study Investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Post-prandial AUC120 | 3 hours from start of meal
  3-hour post-prandial (PP) area under the curve >120 mg/dL (AUC120)

SECONDARY OUTCOMES:
AUC >140 mg/dL | 3 hours from start of meal
  AUC >140 mg/dL over 3 hours PP
Excursion from baseline glucose to peak glucose | 3 hours from start of meal
  Excursion from baseline blood glucose to peak blood glucose during 3 hours PP
Maximum peak glucose | 3 hours from start of meal
  Maximum peak blood glucose during 3 hours PP
Time to peak glucose | 3 hours from start of meal
  Time to peak blood glucose during 3 hours PP
Nadir glucose | 3 hours from start of meal
  Nadir (lowest) blood glucose during 3 hours PP
Mean CGM glucose | 3 hours from start of meal
  Mean CGM glucose during 3 hours PP
Time with glucose >120 mg/dL | 3 hours from start of meal
  Time with blood glucose >120 mg/dL during 3 hours PP
Time with glucose >140 mg/dL | 3 hours from start of meal
  Time with blood glucose >140 mg/dL during 3 hours PP
Glucose ≤140 mg/dL | 1 hour from start of meal
  Blood Glucose ≤140 mg/dL at 1 hour PP
Glucose ≤140 mg/dL | 2 hours from start of meal
  Blood Glucose ≤140 mg/dL at 2 hours PP
Glucose ≤140 mg/dL | 3 hours from start of meal
  Blood Glucose ≤140 mg/dL at 3 hours PP
Glucose ≤120 mg/dL | 1 hour from start of meal
  Blood Glucose ≤120 mg/dL at 1 hour PP
Glucose ≤120 mg/dL | 2 hours from start of meal
  Blood Glucose ≤120 mg/dL at 2 hours PP
Glucose ≤120 mg/dL | 3 hours from start of meal
  Blood Glucose ≤120 mg/dL at 3 hours PP
Time with Glucose in range 63-120 mg/dL | 3 hours from start of meal
  Time with Blood Glucose in range 63-120 mg/dL during 3 hours PP
Time with Glucose in range 63-140 mg/dL | 3 hours from start of meal
  Time with Blood Glucose in range 63-140 mg/dL during 3 hours PP

OTHER OUTCOMES:
Any blood glucose <54 mg/dL | 3 hours from start of meal
  Any blood glucose <54 mg/dL during 3 hours PP
Any blood glucose <63 mg/dL | 3 hours from start of meal
  Any blood glucose <63 mg/dL during 3 hours PP
Any blood glucose <70 mg/dL | 3 hours from start of meal
  Any blood glucose <70 mg/dL during 3 hours PP
Percent time glucose <63 mg/dL | 3 hours from start of meal
  CGM time with glucose <63 mg/dL during 3 hours PP
Hypersensitivity to inhaled technosphere insulin | From the time of administration of the first Technosphere Insulin (TI) dose during the meal session until the end of the calendar day (11:59 PM) on the day of the TI meal session, assessed for up to 18 hours.
  Hypersensitivity reaction, acute bronchospasm, treatment provided for asthma symptoms, or other symptoms associated with TI dosing
Severe Hypoglycemia events during the clinic meal session | From the time of administration of insulin (either Technosphere Insulin [TI] or RAA, depending on the meal session visit) until discharge from the clinic, assessed up to 5 hours for each meal session.
  Any severe hypoglycemia events during the clinic meal session, defined as events requiring assistance of another person due to cognitive impairment to actively administer carbohydrate, glucagon, or other resuscitative actions
Severe hypoglycemia events during the study period | From Screening to Study Completion, an average of 10 days
  Any severe hypoglycemia events during the study period (defined as the time between screening and the final study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Valent, DO, Study Chair — Oregon Health and Science University
Locations (5):
- United States (5):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No